CLINICAL TRIAL: NCT02469441
Title: Does Coffee Intake Reduce Postoperative Ileus After Elective Colorectal Surgery - a Prospective, Randomized Controlled Study - the COFFEE STUDY
Brief Title: Does Coffee Intake Reduce Postoperative Ileus After Elective Colorectal Surgery
Acronym: COFFEE
Status: Completed | Type: Observational
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Gehrer Simone, Dr. med., Kantonsspital Baden
Other Study IDs: 2014-062
Record Dates: First submitted 2015-05-29; First posted 2015-06-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Ileus
Keywords: coffee; postoperative ileus; colorectal surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arm A: Arm A (treatment arm: coffee): patients after colorectal surgery receive coffee in addition to the regular infusion therapy and/or alimentation
- Arm B: Arm B (control arm: water / tea): patients after colorectal surgery receive water or tea (excluding black tea) and no coffee until the first bowel movement in addition to the regular infusion therapy and/or alimentation

SUMMARY:
The aim of the study is to investigate if postoperative coffee intake decreases the time until first bowel movement in elective colorectal surgery with primary anastomosis.

DETAILED DESCRIPTION:
Postoperative ileus after colorectal surgery is a frequent problem which significantly prolongs hospital stay and increases perioperative costs. Postoperative therapeutic interventions vary significantly between different hospitals due to missing evidence-based guidelines. Coffee is a safe, cheap and simple agent without significant side effects which can positively influence the bowel function.

The aim of the investigators is to evaluate in an own study if coffee consumption has an influence on the duration of postoperative ileus.

The present trial is designed to evaluate if postoperative coffee intake decreases the time until first bowel movement in colorectal surgery with primary anastomosis. This study would be the second study which evaluates the described questions under randomized conditions.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for elective laparoscopic or open colorectal surgery due to benign or malignant colorectal disease, which need a large bowel resection with primary anastomosis

* Age equal or greater than 18 years
* Patients that are able to give informed consent
* Elective Surgery
* Anastomosis above 6 cm from anal verge

Exclusion Criteria:

* Participation in other studies
* Additional small bowel anastomosis
* Need for extended adhesiolysis
* Need for a stoma (e.g. protective ileostomy)
* Emergency operation with diffuse peritonitis or preexisting ileus
* Preoperative radiation
* Known hypersensitivity or allergy to coffee
* Expected lack of compliance
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with elective colorectal surgery and primary anastomosis > 6cm above the anal verge without stoma formation
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Time to first bowel movement | Follow-up per patient: 1 month postoperatively
  Time to first bowel movement (time from the end of surgery until the first passage of stool recorded by nursing staff) as a marker for the termination of postoperative ileus.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Hasler-Gehrer, MD, Principal Investigator — Oberärztin
Locations (1):
- Kantonsspital Baden, Baden, Switzerland

REFERENCES:
- [Derived] Hasler-Gehrer S, Linecker M, Keerl A, Slieker J, Descloux A, Rosenberg R, Seifert B, Nocito A. Does Coffee Intake Reduce Postoperative Ileus After Laparoscopic Elective Colorectal Surgery? A Prospective, Randomized Controlled Study: The Coffee Study. Dis Colon Rectum. 2019 Aug;62(8):997-1004. doi: 10.1097/DCR.0000000000001405. PMID 30998528